CLINICAL TRIAL: NCT04256577
Title: Serum Ceramides Level in Systemic Lupus Erythematosus (SLE) Patients as a Novel Marker for Renal Impairment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, NADIA HUSSIEN HAMMAM HUSSIEN, resident doctor, Assiut University
Other Study IDs: serum ceramides level in (SLE)
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-01

CONDITIONS: Systemic Lupus
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients proven having (SLE): 20 patients proven to have systemic lupus Erthematosus without renal impairment (eGFR) ≥ 80 ml/min/1.73 m2 and albumin / creatinine ≤ 30 mg/g)
  Interventions: Diagnostic Test: serum ceramides level in blood
- patients proven to have (LN) by renal biopsy: Group (2) 25 patients proven to have LN by renal biopsy before starting treatment and after 3 cycle of treatment (eGFR < 80 ml/min/1.73 m2 and albumin/creatinine ratio > 30 mg/g)
  Interventions: Diagnostic Test: serum ceramides level in blood
- healthy control: (20) patients healthy control matched in age and sex
  Interventions: Diagnostic Test: serum ceramides level in blood

INTERVENTIONS:
Diagnostic Test: serum ceramides level in blood — Serum ceramides ( sphingolipid measurement, plasma (EDTA as anticoagulant) and serum separation was performed immediately after blood drawing by two-time scentrifugation at 750 x g for 5 min (4°C). Lipid extraction from plasma and/or serum samples (10 µl each) and subsequent LC-MS/MS)

SUMMARY:
1. Estimation of serum ceramides level in SLE patients as anovel marker for renal impairment
2. Correlation serum ceramides level with histological classification of LN,C3,C4,ANA,ANTI DS DNA ,CRP ,ESR , eGFR , creatinine /protein ratio
3. Follow up estimation of ceramides level in LN patients after 3 cycles of treatment

DETAILED DESCRIPTION:
Systemic lupus erythrematosus (SLE) is an autoimmune disease with increasing prevalence and incidence , The clinical manifestation is multifaceted and targets the musculoskeletal system, the skin and different organs like lung and kidney From 30-80% of SLE patients develop lupus nephritis (LN) which often leads to chronic kidney disease (CKD) and end-stage renal disease (ESRD) and is associated with an overall poor prognosis and high mortality Diagnosis of LN is made by kidney biopsy, which still remains the gold standard Histological evaluation distinguish between different stages of LN upon morphological changes within the kidney . However, noninvasive methods to diagnose and guide LN therapy are currently not established in the clinic. On the other hand, an early diagnosis is important for the therapeutic success and thereby lowers the risk of ESRD In this context, classical clinical markers for renal dysfunction are insufficient for an early assessment of the need for renal biopsies and subsequently to decide about the optimal therapy. Even though traditional biomarkers like antids DNA antibodies and complement deficiency are widely accepted as diagnostic instruments to assess disease activity, their specificity is rather low, and they appear to be more suitable to confirm diagnosis of SLE and LN in an already likely clinical setting Ceramides are a family of waxy lipid molecules ,composed of sphingosine and fatty acide ,found in high concentration with in the cell membrane of eukaryocyte cells, since they are component lipids that make up sphingomyelin, one of the major lipids in the lipid bilayer Ceramides and other sphingolipids found in cell membrane were purely supporting structural elements,also participate in variety of cellular signaling, regulating differentiation, proliferation, Programmed cell death(PCD) Sphingolipids are a heterogenous group of lipids with more than 400 single compounds formed by structural and chemical modifications of a sphingosine backbone Recent studies reveal that blood sphingolipids not only have important signaling properties but also serve as biomarkers in various renal disease Patyna etal in 2019 concluded that ceramides in blood could act as potent biomarker for renal impairment in patient

ELIGIBILITY:
Inclusion Criteria:

* Forty five patients will SLE with and without renal impairment diagnosed as SLE according to SLICC classification criteria for SLE

Exclusion Criteria:

* Malignant tumor ,infectious diseases, Alzheimer disease ,type 2 diabetes mellitus vitamin D intaker, obesty , cardiovascular disease (HTN,HF ,ischemic heart disease)

Ages: 17 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Prospective analytic (cross_section) study will be carried out on patients admitted to assiut university hospital internal medicine department.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Estimation of serum ceramides level in SLE patients as anovel marker for renal impairment | base line
  Correlation serum ceramides level with histological classification of LN,C3,C4,ANA,ANTI DS DNA ,CRP ,ESR , eGFR , creatinine /protein ratio

REFERENCES:
- [Background] Patyna S, Buttner S, Eckes T, Obermuller N, Bartel C, Braner A, Trautmann S, Thomas D, Geiger H, Pfeilschifter J, Koch A. Blood ceramides as novel markers for renal impairment in systemic lupus erythematosus. Prostaglandins Other Lipid Mediat. 2019 Oct;144:106348. doi: 10.1016/j.prostaglandins.2019.106348. Epub 2019 Jul 10. PMID 31301404